CLINICAL TRIAL: NCT02790229
Title: Outcome of Patients After Lower Limb Fracture With Partial Weight Bearing Postoperatively Treated With or Without Anti-gravity Treadmill (Alter G®) During Six Weeks of Rehabilitation - a Bicentric Prospective Randomized Trial
Brief Title: Postoperatively Treated Patients With Lower Limb Fracture With or Without an Anti-gravity Treadmill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Ambulantes Reha Centrum Gruppe, Germany (Unknown); Hospital St.Georg gGmbH; Clinic of Trauma, Orthopedic and septic Surgery, Leipzig, Germany (Unknown)
Responsible Party: Principal Investigator, Dr. med. Ralf Henkelmann, Dr. med. Ralf Henkelmann, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR-0244
Record Dates: First submitted 2016-05-29; First posted 2016-06-03 (Estimated); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Muscle Degeneration
Keywords: rehabilitation, anti-gravity treadmill

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anti-gravity treadmill arm (Experimental): Treatment with anti-gravity treadmill (alter G®)
  Interventions: Other: anti-gravity treadmill (alter G®)
- control arm (Other): Treatment with standardized physiotherapy
  Interventions: Other: standardized physiotherapy

INTERVENTIONS:
Other: anti-gravity treadmill (alter G®) — Patients in the experimental arm will be treated with manual lymphatic drainage, cryotherapy and a fixed protocol of training in an anti-gravity treadmill (alter G®). The protocol is designed parallel to standard physiotherapy with a frequency of two to three times a week with duration of about 20 minutes for six weeks.
  Arms: anti-gravity treadmill arm
Other: standardized physiotherapy — Patients in the control arm will be treated with manual lymphatic drainage, cryotherapy and 20 minutes of physiotherapy two to three times a week for six weeks. Physiotherapy will be done according to a standardized protocol.
  Arms: control arm

SUMMARY:
The presented study is designed to prove efficacy of the anti-gravity treadmill (alter G®) compared to a standard rehabilitation protocol in patients with tibial plateau or ankle fractures with six weeks of partial weight bearing.

ELIGIBILITY:
Inclusion Criteria:

* patients with a postoperative partial weight bearing after tibial plateau or ankle fracture.
* man and woman of an age between 18 and 65

Exclusion Criteria:

* Body weight more than 100kg
* serious illness or poor general health as judged by physician that may influence the rehabilitation
* open fractures (>1° according to Gustilo and Anderson)
* surgical site infection
* pregnancy
* neuromuscular disorders or preexisting muscle atrophy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-08; Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Change of overall KOOS or FOAS | 12 months
  Change of overall KOOS (Knee Injury and Osteoarthritis Outcome Score) or FOAS (Foot and Ankle Outcome Score) from baseline (Day 1 after operation) to Final Assessment (FA) 12 months after operation determined for each group and between the groups.

SECONDARY OUTCOMES:
Change of the 5 subscores of the KOOS or FAOS | Baseline to 6 and 12 weeks and 12 months
  Change of the 5 subscores of the KOOS or FAOS (Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec), knee/ankle related Quality of life (QoL)) determined for each group and between the groups.
Circumference measurement of tights and lower leg on both legs | Baseline to day of discharge, 3,6 and 12 weeks and 12 months
  Circumference measurement of tights and lower leg on both legs 10cm and 20cm above the knee joint space and 10cm below (knee in neutral position) from baseline (Day 1 after operation) to day of discharge (7-11d), 3, 6 and 12 weeks and 12 months (FA) after operation determined for each group and between the groups.
ROM | Baseline to 6 and 12 weeks and 12 months
  Range of motion (ROM) of the affected joint determined by neutral zero method from baseline (Day 1 after operation) to 6 and 12 weeks and 12 months after operation determined for each group and between the groups.
SF-36 | Baseline to 6 and 12 weeks and 12 months
  Short Form Health Survey (SF-36) from baseline (Day 1 after operation) to 6 and 12 weeks and 12 months after operation determined for each group and between the groups.
DGI | day of discharge to 3, 6 and 12 weeks and 12 months postoperative
  Dynamic gait index (DGI) from day of discharge (7-11d) to 3, 6 and 12 weeks and 12 months after operation determined for each group and between the groups.

OTHER OUTCOMES:
Absence from work | 12 months
  Number of days of absence from work (employment) and/or days of inability to follow usual activities until FA and time point when patient was back to work and/or to follow usual activities. Data recorded for each group and compared between the groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Leipzig, Clinic of Orthopedic, Trauma and Plastic Surgery, Leipzig, Saxony
  - Klinikum St. Georg gGmbH, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Webber SC, Horvey KJ, Yurach Pikaluk MT, Butcher SJ. Cardiovascular responses in older adults with total knee arthroplasty at rest and with exercise on a positive pressure treadmill. Eur J Appl Physiol. 2014 Mar;114(3):653-62. doi: 10.1007/s00421-013-2798-1. Epub 2013 Dec 22. PMID 24362964
- [Background] Suetta C, Frandsen U, Mackey AL, Jensen L, Hvid LG, Bayer ML, Petersson SJ, Schroder HD, Andersen JL, Aagaard P, Schjerling P, Kjaer M. Ageing is associated with diminished muscle re-growth and myogenic precursor cell expansion early after immobility-induced atrophy in human skeletal muscle. J Physiol. 2013 Aug 1;591(15):3789-804. doi: 10.1113/jphysiol.2013.257121. Epub 2013 Jun 3. PMID 23732643
- [Background] Saxena A, Granot A. Use of an anti-gravity treadmill in the rehabilitation of the operated achilles tendon: a pilot study. J Foot Ankle Surg. 2011 Sep-Oct;50(5):558-61. doi: 10.1053/j.jfas.2011.04.045. Epub 2011 Jun 23. PMID 21703879
- [Background] Takacs J, Leiter JR, Peeler JD. Novel application of lower body positive-pressure in the rehabilitation of an individual with multiple lower extremity fractures. J Rehabil Med. 2011 Jun;43(7):653-6. doi: 10.2340/16501977-0806. PMID 21584484
- [Background] Peeler J, Christian M, Cooper J, Leiter J, MacDonald P. Managing Knee Osteoarthritis: The Effects of Body Weight Supported Physical Activity on Joint Pain, Function, and Thigh Muscle Strength. Clin J Sport Med. 2015 Nov;25(6):518-23. doi: 10.1097/JSM.0000000000000173. PMID 25647537
- [Background] Moore MN, Vandenakker-Albanese C, Hoffman MD. Use of partial body-weight support for aggressive return to running after lumbar disk herniation: a case report. Arch Phys Med Rehabil. 2010 May;91(5):803-5. doi: 10.1016/j.apmr.2010.01.014. PMID 20434621
- [Background] McNeill DK, de Heer HD, Bounds RG, Coast JR. Accuracy of unloading with the anti-gravity treadmill. J Strength Cond Res. 2015 Mar;29(3):863-8. doi: 10.1519/JSC.0000000000000678. PMID 25226319
- [Background] Hoffman MD, Donaghe HE. Physiological responses to body weight--supported treadmill exercise in healthy adults. Arch Phys Med Rehabil. 2011 Jun;92(6):960-6. doi: 10.1016/j.apmr.2010.12.035. PMID 21621673
- [Background] Cutuk A, Groppo ER, Quigley EJ, White KW, Pedowitz RA, Hargens AR. Ambulation in simulated fractional gravity using lower body positive pressure: cardiovascular safety and gait analyses. J Appl Physiol (1985). 2006 Sep;101(3):771-7. doi: 10.1152/japplphysiol.00644.2005. Epub 2006 Jun 15. PMID 16777997
- [Derived] Henkelmann R, Schneider S, Muller D, Gahr R, Josten C, Bohme J. Outcome of patients after lower limb fracture with partial weight bearing postoperatively treated with or without anti-gravity treadmill (alter G(R)) during six weeks of rehabilitation - a protocol of a prospective randomized trial. BMC Musculoskelet Disord. 2017 Mar 14;18(1):104. doi: 10.1186/s12891-017-1461-0. PMID 28288613